CLINICAL TRIAL: NCT00778011
Title: Ondansetron 4 mg vs. 2 mg vs. Metoclopramide 10 mg for Nausea and Vomiting in the Emergency Department: A Randomized, Double-Blind Clinical Trial
Brief Title: Uncomplicated Nausea and Vomiting in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Marc Pollack, MD, PhD, York Hospital Emergency Medicine Physician
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0506018
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Ondansetron; Metoclopramide; Randomized; Double-Blind; nausea and vomiting in the emergency department
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Ondansetron
- 2 (Active Comparator)
  Interventions: Drug: Ondansetron
- 3 (Active Comparator)
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Ondansetron — dosage
  Other Names: Ondansetron 2 mg IV
  Arms: 1
Drug: Ondansetron — 4 mg
  Other Names: Ondansetron 4 mg IV
  Arms: 2
Drug: Metoclopramide — 10 mg IV
  Other Names: Metoclopramide 10 mg IV
  Arms: 3

SUMMARY:
Nausea and vomiting is a common complaint in the emergency department. Treatment is important for many reasons. In addition to patient comfort, there are adverse effects secondary to vomiting such as dehydration, metabolic alkalosis, Mallory-Weiss tears, and aspiration. Two mediations common used for nausea in ED patients include Ondanesetron and Metoclopramide.

DETAILED DESCRIPTION:
This study will compare Ondansetron 4 mg vs 2 mg vs Metoclopramide 10 mg to look for efficacy in nausea and vomiting treatment for patients in the ED with many different causes. We will also look for cost effectiveness as well, since Metoclopramide is much less expensive than Ondansetron, which is less expensive at lower doses. There is little research about nausea medication in the ED literature even though these medications are used frequently in the ED for many causes of nausea.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with nausea and at least 1 episode vomiting in the last 12 hours presenting to the York Hospital Emergency Department

Exclusion Criteria:

* Patients known to have hypersensitivity to the drugs ondansetron or metoclopramide
* gastrointestinal hemorrhage, mechanical obstruction or perforation
* patients with pheochromocytoma
* seizure disorder
* patients receiving other drugs which are likely to cause extrapyramidal reactions such as butapherones and phenothiazines
* patients experiencing hyperemesis gravidum
* patients unable to understand the informed consent (intoxicated, Spanish speaking)
* prior antiemetics within 12 hours
* inability to perform visual analog scale
* renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To delineate whether a high vs low dose of Ondansetron in better as opposed to an alternate medication -- Metoclopramide in the ED setting for uncomplicated nausea and vomiting. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pollack, MD, PhD, Principal Investigator — York Hospital Emergency Department Physician
Locations (1):
- York Hospital, York, Pennsylvania, United States